CLINICAL TRIAL: NCT01011699
Title: Comparison of Nicotinamide and Sevelamer Hydrochloride on Phosphatemia Control on Chronic Hemodialysed Patients
Brief Title: Nicotinamide Versus Sevelamer Hydrochloride on Phosphatemia Control on Chronic Hemodialysed Patients
Acronym: NICOREN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Financial problem
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PHRCIR08-PR-FOURNIER; Eudract N°2008-004673-17 (Other: AFSSAPS)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Renal Failure; Hemodialysis
Keywords: nicotinamide; sevelamer hydrochloride; phosphatemia; cinacalcet; dyslipidemia; vascular calcification; bone mass loss
MeSH Terms: conditions — Kidney Failure, Chronic; Dyslipidemias; Vascular Calcification | interventions — Niacinamide; Sevelamer; Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevelamer (Active Comparator): Titration phase with sevelamer (Renagel) with the aim of phosphatemia control in 4 weeks of treatment, with stable dose of calcic carbonate.
  Increase of sevelamer dose up to 12 tablets, as follows:
  0 morning, 2 noon, 2 evening (first week), then, 0 morning, 4 noon, 4 evening (second week), then, 2 morning, 4 noon, 4 evening (third week), then, 4 morning, 4 noon, 4 evening (fourth week).
  Interventions: Drug: sevelamer; Drug: cinacalcet
- nicotinamide (Active Comparator): Titration phase with nicotinamide (Nicobion) with the aim of phosphatemia control in 4 weeks of treatment, with stable dose of calcic carbonate.
  Increase of nicotinamide dose up to 4 tablets, as follows:
  0 morning, 1 noon, 0 evening (first week), then, 0 morning, 1 noon, 1 evening (second week), then, 1 morning, 1 noon, 1 evening (third week), then, 1 morning, 2 noon, 1 evening (fourth week).
  Interventions: Drug: nicotinamide; Drug: cinacalcet

INTERVENTIONS:
Drug: nicotinamide — Titration phase of nicotinamide (Nicobion) with the aim of phosphatemia control in 4 weeks with stable dose of calcic carbonate;
  Increase of nicotinamide dose of Nicobion 500mg (nicotinamide 500mg), up to 4 tablets daily, as follows:
  0 morning, 1 noon, 0 evening (first week), then, 0 morning, 1 noon, 1 evening (second week), then, 1 morning, 1 noon, 1 evening (third week), then, 1 morning, 2 noon, 1 evening (fourth week).
  Other Names: Nicobion; ATC class A11HA01
  Arms: nicotinamide
Drug: sevelamer — Titration phase with sevelamer (Renagel) with the aim of phosphatemia control before 4 weeks of treatment, with stable dose of calcic carbonate.
  Increase of sevelamer dose up to 12 tablets, as follows:
  0 morning, 2 noon, 2 evening (first week), then, 0 morning, 4 noon, 4 evening (second week), then, 2 morning, 4 noon, 4 evening (third week), then, 4 morning, 4 noon, 4 evening (fourth week).
  Other Names: Renagel; ATC class V03AE02
  Arms: sevelamer
Drug: cinacalcet — After 6 months of treatment, patient screening on PTH level:
  For patients with PTH > 300pg/ml, introduction of cinacalcet by level of 30 mg every 3 weeks, up to 180mg daily (administered during the meal and before next dialysis) Cinacalcet increase will be stopped once PTH < 250 pg/ml. Calcic carbonate dose will be increase once calcemia will be < 2.25 mmol/l. If maximum tolerated dose is not sufficient to prevent hypocalcemia < 2.10 mmol/l calcium of dialysis bath wille be increased up to 1.75 mmol/l and calcic carbonate will be decreased.
  A dose adjustment is possible with nicotinamide to obtain a phosphatemia between 1.10 and 1.60 mmol/l.
  Other Names: Mimpara; ATC class H05BX01

SUMMARY:
The comparison between nicotinamide and sevelamer aims to demonstrate, in chronic hemodialysed patients, the non-inferiority of nicotinamide in terms of control of the phosphatemia. Secondary objectives is to compare the two treatments in terms of efficiency in other biological parameters, vascular calcification and bone mass loss and on the clinical and biological tolerance and finally to explore the roles of metabolites of nicotinamide.

DETAILED DESCRIPTION:
This is a multicenter randomized open study with 2 treatment arms (nicotinamide / Sevelamer).

Laboratories who will dose biochemical parameters and PTH, ignore which treatment is received by patients.

The team which will measure bone density and the radiologist or rheumatologist who will appreciate centrally calcification and deformity of the vertebrae, ignore which treatment is received by patients.

Therefore it's a Randomized Prospective Blinded Outcome Endpoint.

Pre-recruitment period (3 to 6 months) with basic medication

* Repletion of vitamin D (p 25 OHD between 30 and 50 ng / ml) (if required by supplementation Dedrogyl weekly by the dialysis nurse)
* Bath dialysis to 1.50 mmol / l calcium (1.75 mmol / l if hemodiafiltration), 32 mmol bicarbonate and 0.5 mmol / l magnesium - Support to provide a dietary protein intake with 1.2 g / kg / d and assessment of contributions of Ca and PO4
* Use of CaCO3 taken with meals rich in phosphorus (morning, noon and evening) without
* In case of hyperkalemia, Calcium Sorbisterit® will preferably be used instead of KAYEXALATE®. This process exposes the worsening effect of hyperphosphatemia increasing calcium malabsorption and therefore the negative calcium balance in renal failure.
* Statin therapy, fibrate or ezetimibe if necessary, but with stable dose

This treatment will be monitored on the following parameters:

* Biochemical weekly Predialytic (midweek): creatinine, urea, PO4, Ca, protein, Na, K, bicarbonate, glucose, uric acid
* Additional monthly balance: PTH intact, Mg, albumin, CRP
* Each 4 months update: lipid profile (fasting or not, but always at the same time, 25 OH D, complete blood count (CBC), AST-ALT, total alkaline phosphatase, gamma-GT, PKC, glycated hemoglobin (HbA1C) )

Recruitment (180 patients):

* Obtaining informed consent
* Perform a bone density by DXA third of the radius (cortical bone), radius ultradistal (trabecular bone), femoral neck bone (mixed), whole body and lumbar spine profile radiography.
* Lumbar and dorsal radiography (frontal and profile) for research and vertebral measurement of aortic calcification by the Framingham score) + pelvis radiography (frontal) and 2 hands radiography (frontal) searching vascular calcification, Looser's streaks and subperiosteal resorption.
* Freezing at -80 ° C (4 tubes of 1 ml of serum)for centralized analysis:PTH, 25 OHD, CTX, PAO. All samples will be sent for laboratory analysis of Biochemistry University Hospital of Amiens at the end of the study.

For this, 10 ml of blood will be collected with a dry tube then centrifuged 15 minutes, 4000-5000 rpm at room temperature within 30 minutes after collection. Then, aliquot 1ml into 4 polypropylene tubes being careful not to take the fibrin.

* Freezing at -80 ° C in a tube of 2.5 ml of plasma to be assayed later the metabolites of nicotinamide. These samples will only be achieved if patients accept and mark the second part of the consent. The tubes are then stored in the biological resource center, CHU Amiens for further research and for an indefinite period.

The nicotinamide metabolites measured in this study will annex the Met2PY (N-methyl-2-pyridone-5-carboxamide), the Met4PY (N-methyl-4-pyridone-3-carboxamide) and NAD (nicotinamide adenine dinucleotide).

6 ml of EDTA whole blood will be collected, then centrifuged 15 minutes, 4000-5000 rpm at room temperature within 30 minutes after collection. Then, 2.5 ml aliquot in 1 polypropylene tube.

* Then a heparinized blood sample of 2.5 ml will be frozen at -80 °C for determination of nicotinamide. All samples will be sent for analysis at CERBA at the end of the study.

Randomization will be done by the minimization technic with stratification factors: center, duration of dialysis and taking lipid lowering therapy. Randomization will be performed remotely via a website.

Follow-up of one year:

* Period titration nicotinamide or sevelamer to control serum phosphorus in 4 weeks, with stable doses of CaCO3
* Increased nicotinamide 500 mg up to 4 tablets: 0-1-0, 0-1-1, 1-1-1, 1-2-1
* Increased sevelamer 800 mg up to 12 tablets: 0-2-2 ; 2-4-4 ; 4-4-4 ; 2-5-5
* Maintenance period of 5 months with assessment of maintenance doses of Renagel (sevelamer) or Nicobion (nicotinamide) or during the last 3 months.
* After these 6 months:
* Freezing -80 ° C, 4 tubes of 1 ml of serum centralized reviews PTH, 25 OHD, CTX, PAO (as mentioned above).
* Freezing -80 ° C in a tube of 2.5 ml of plasma to be assayed later the metabolites of nicotinamide (as mentioned above).
* Freezing -80 ° C with a heparinized blood sample of 2.5 ml for determination of nicotinamide (as mentioned above).
* Second randomization via a website, patients with intact PTH> 300 pg / ml after 6 months of Nicobion ® and Renagel ®. Randomization 75-150 pg / ml or 150-300 mg / ml will be made by the minimization technic with stratification factors: the center and the type of Hypophosphatemia PTH will be reduced by introducing cinacalcet ® by increments of 30 mg every 3 weeks to 180 mg / day (given with meals 24 hours before the next dialysis). Increase of Cinacalcet ® will be stopped when PTH is <250 pg / ml for arm 150-300pg/ml or <125 per arm 75-150 pg / ml.

Once corrected calcemia <2.25 mmol / l, doses of CaCO3 will be increased; if the maximum tolerable of CaCO3 on the tract map does not prevent hypocalcemia (<2.10 mmol / l), the calcium bath will be increased to 1.75 mmol / l CaCO3 decreased and, if necessary adjustment of nicotinamide / Sevelamer to maintain PO4 between 1.30 and 1.60 mmol / l.

* During the first 6 months of administration of sevelamer, weekly, monthly and quarterly reports will be done. Regarding PTH assay will be performed, every 3 weeks during the titration of cinacalcet.
* A lumbar and dorsal radiography (frontal and profile), a pelvis radiography (face) and 2 hands radiography (front) will be conducted at the end of follow-up period.
* Bone densitometry will be performed at the end of the study (same camera - same site).
* Case report form: tolerance, serious adverse events, compliance, cardiovascular events (myocardial infarction, PAO, stroke, arteritis, vascular intervention),deaths and fractures during the follow-up study.
* Freezing -80 ° C to 4 tubes of 1 ml of serum centralized reviews PTH, 25 OHD, CTX, PAO at the end of the study (as mentioned above).
* Freezing -80 ° C in a tube of 2.5 ml of plasma to be assayed later the metabolites of nicotinamide at the end of the study (as mentioned above).
* Freezing at -80 ° C with a heparinized blood sample of 2.5 ml for determination of nicotinamide at the end of the study (as mentioned above).

Analytical Methodology

ELIGIBILITY:
Inclusion Criteria:

* Women or men over 18 years
* Chronic hemodialysis (since more than 3 months)
* Hyperphosphatemia controlled with only CaCO3
* PO4 > 1,60 mmol/l, PCa < 2,37 mmol/l
* patient able to understand and sign informed consent form

Exclusion Criteria:

* PTH < 60 ou > 800 pg/ml (PTX)
* Aluminium intoxication (aluminium level in blood > 0,5 µmol/l)
* Score of aortic calcifications ≥ 20 (max 24)
* Characterized intolerance with Renagel and/or Nicobion
* Pregnant woman
* Autoimmune disease
* Patient known to have a bad drug compliance
* Blood tests abnormality (thrombopenia <150 000, serum albumin <30g)
* Hepatic tests abnormality
* Transplant probably within 6 months
* Patient who will need transplantation within 6 month
* Patients receiving chemotherapy
* Patients having a loss of dry weight of 3 kg in 3 months or 6 kg in 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The comparison between nicotinamide and Sevelamer was primarily to demonstrate the noninferiority of nicotinamide in terms of control of the phosphatemia observed during the 4th, 5th and 6th months before to introduce Cinacalcet ®. | 6th months

SECONDARY OUTCOMES:
To demonstrate noninferiority of nicotinamide in terms of effect on dyslipidemia (evaluated by the ratio LDL / HDL cholesterol), the risk of hypercalcemia (PCa> 2.37 mmol / l) and increase of phospho-calcic product (> 3 , 79 mmol/l). | 6 th months and one year
To evaluate the difference between nicotinamide and sevelamer on vascular calcification | one year
To evaluate the difference between nicotinamide and sevelamer on bone mass loss and fracture risk | one year
Evaluate the percentage of population requiring use of cinacalcet® to control PTH (75-300 pg/ml). Evaluate his benefit on phosphatemia and calcemia control. Prevent the need for surgical PTX, and evaluate the additional cost of treatment by cinacalcet | 6th months
Evaluate roles of metabolites of nicotinamide (efficacy and side effects) through another study | 6th months and one year
Compare the cost-effectiveness ratio of these two treatments | one year

CONTACTS AND LOCATIONS:
Overall Officials: Albert FOURNIER, Pr, Study Director — Centre Hospitalier Universitaire, Amiens; Ziad MASSY, Pr, Principal Investigator — Centre Hospitalier Universitaire, Amiens
Locations (18):
- France (18):
  - Centre Hospitalier Général, Soissons, Aisne
  - Centre Hospitalier, Lisieux, Calvados
  - Centre Hospitalier, Cambrai, Cambrai
  - Association pour le Développement de l'Hémodialyse, Hénin-Beaumont, Hauts-de-France
  - ALURAD, Limoges, Limousin
  - Centre Hospitalier Universitaire, Reims, Marne
  - Association Régionale Promotion Dialyse à domicile (ARPDD), Reims, Marne
  - Polyclinique de la Louvière, Lille, Nord
  - CHRU, Lille, Nord
  - Hôpital Victor Provo, Roubaix, Nord
  - Centre Hospitalier Général, Valenciennes, Nord
  - Centre Hospitalier Général, Beauvais, Oise
  - Clinique Saint Côme, Compiègne, Oise
  - Centre Hospitalier Général, Creil, Oise
  - Clinique du Bois Bernard, Bois-Bernard, Pas de calais
  - Centre Hospitalier, Boulogne-sur-Mer, Pas de calais
  - Centre Hospital-Universitaire d'Amiens, Amiens, Picardie
  - Clinique de l'Europe, Rouen, Seine maritime

REFERENCES:
- [Background] Goldsmith D, Ritz E, Covic A. Vascular calcification: a stiff challenge for the nephrologist: does preventing bone disease cause arterial disease? Kidney Int. 2004 Oct;66(4):1315-33. doi: 10.1111/j.1523-1755.2004.00895.x. PMID 15458425
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Epidemiology of cardiovascular disease in chronic renal disease. J Am Soc Nephrol. 1998 Dec;9(12 Suppl):S16-23. PMID 11443763
- [Background] K/DOQI: (Kidney Disease Outcomes Quality Initiative) of the National Kidney Foundation. Am J Kidney Dis suppl 3, october 2003.
- [Background] Jungers P, Choukroun G, Robino C, Massy ZA, Taupin P, Labrunie M, Man NK, Landais P. Epidemiology of end-stage renal disease in the Ile-de-France area: a prospective study in 1998. Nephrol Dial Transplant. 2000 Dec;15(12):2000-6. doi: 10.1093/ndt/15.12.2000. PMID 11096146
- [Background] Kalantar-Zadeh K, Block G, Humphreys MH, Kopple JD. Reverse epidemiology of cardiovascular risk factors in maintenance dialysis patients. Kidney Int. 2003 Mar;63(3):793-808. doi: 10.1046/j.1523-1755.2003.00803.x. PMID 12631061
- [Background] Collins R, Armitage J, Parish S, Sleigh P, Peto R; Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol-lowering with simvastatin in 5963 people with diabetes: a randomised placebo-controlled trial. Lancet. 2003 Jun 14;361(9374):2005-16. doi: 10.1016/s0140-6736(03)13636-7. PMID 12814710
- [Background] London GM, Guerin AP, Marchais SJ, Metivier F, Pannier B, Adda H. Arterial media calcification in end-stage renal disease: impact on all-cause and cardiovascular mortality. Nephrol Dial Transplant. 2003 Sep;18(9):1731-40. doi: 10.1093/ndt/gfg414. PMID 12937218
- [Background] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Background] Shahapuni I, Mansour J, Harbouche L, Maouad B, Benyahia M, Rahmouni K, Oprisiu R, Bonne JF, Monge M, El Esper N, Presne C, Moriniere P, Choukroun G, Fournier A. How do calcimimetics fit into the management of parathyroid hormone, calcium, and phosphate disturbances in dialysis patients? Semin Dial. 2005 May-Jun;18(3):226-38. doi: 10.1111/j.1525-139X.2005.18318.x. PMID 15934970
- [Background] Ghazali A, Fardellone P, Pruna A, Atik A, Achard JM, Oprisiu R, Brazier M, Remond A, Moriniere P, Garabedian M, Eastwood J, Fournier A. Is low plasma 25-(OH)vitamin D a major risk factor for hyperparathyroidism and Looser's zones independent of calcitriol? Kidney Int. 1999 Jun;55(6):2169-77. doi: 10.1046/j.1523-1755.1999.00480.x. PMID 10354266
- [Background] Goldsmith DJ, Covic A, Sambrook PA, Ackrill P. Vascular calcification in long-term haemodialysis patients in a single unit: a retrospective analysis. Nephron. 1997;77(1):37-43. doi: 10.1159/000190244. PMID 9380236
- [Background] Teng M, Wolf M, Lowrie E, Ofsthun N, Lazarus JM, Thadhani R. Survival of patients undergoing hemodialysis with paricalcitol or calcitriol therapy. N Engl J Med. 2003 Jul 31;349(5):446-56. doi: 10.1056/NEJMoa022536. PMID 12890843
- [Background] Fournier AE, Johnson WJ, Taves DR, Beabout JW, Arnaud CD, Goldsmith RS. Etiology of hyperparathyroidism and bone disease during chronic hemodialysis. I. Association of bone disease with potentially etiologic factors. J Clin Invest. 1971 Mar;50(3):592-8. doi: 10.1172/JCI106529. PMID 5101783
- [Background] Argiles A, Kerr PG, Canaud B, Flavier JL, Mion C. Calcium kinetics and the long-term effects of lowering dialysate calcium concentration. Kidney Int. 1993 Mar;43(3):630-40. doi: 10.1038/ki.1993.92. PMID 8455362
- [Background] Indridason OS, Quarles LD. Comparison of treatments for mild secondary hyperparathyroidism in hemodialysis patients. Durham Renal Osteodystrophy Study Group. Kidney Int. 2000 Jan;57(1):282-92. doi: 10.1046/j.1523-1755.2000.00819.x. PMID 10620210
- [Background] Locatelli F, Covic A, Chazot C, Leunissen K, Luno J, Yaqoob M. Optimal composition of the dialysate, with emphasis on its influence on blood pressure. Nephrol Dial Transplant. 2004 Apr;19(4):785-96. doi: 10.1093/ndt/gfh102. PMID 15031331
- [Background] Chertow GM, Burke SK, Raggi P; Treat to Goal Working Group. Sevelamer attenuates the progression of coronary and aortic calcification in hemodialysis patients. Kidney Int. 2002 Jul;62(1):245-52. doi: 10.1046/j.1523-1755.2002.00434.x. PMID 12081584
- [Background] Fournier A, Said S, Ghazali A, Sechet A, Ezaitouni F, Marie A, Westeel PF, Moriniere P, Boudailliez B. The clinical significance of adynamic bone disease in uremia. Adv Nephrol Necker Hosp. 1997;27:131-66. No abstract available. PMID 9408446
- [Background] London GM, Marty C, Marchais SJ, Guerin AP, Metivier F, de Vernejoul MC. Arterial calcifications and bone histomorphometry in end-stage renal disease. J Am Soc Nephrol. 2004 Jul;15(7):1943-51. doi: 10.1097/01.asn.0000129337.50739.48. PMID 15213285
- [Background] Delmez JA, Tindira CA, Windus DW, Norwood KY, Giles KS, Nighswander TL, Slatopolsky E. Calcium acetate as a phosphorus binder in hemodialysis patients. J Am Soc Nephrol. 1992 Jul;3(1):96-102. doi: 10.1681/ASN.V3196. PMID 1391713
- [Background] Ben Hamida F, el Esper I, Compagnon M, Moriniere P, Fournier A. Long-term (6 months) cross-over comparison of calcium acetate with calcium carbonate as phosphate binder. Nephron. 1993;63(3):258-62. doi: 10.1159/000187207. PMID 8446261
- [Background] Yang H, Curinga G, Giachelli CM. Elevated extracellular calcium levels induce smooth muscle cell matrix mineralization in vitro. Kidney Int. 2004 Dec;66(6):2293-9. doi: 10.1111/j.1523-1755.2004.66015.x. PMID 15569318
- [Background] Porsti I, Fan M, Koobi P, Jolma P, Kalliovalkama J, Vehmas TI, Helin H, Holthofer H, Mervaala E, Nyman T, Tikkanen I. High calcium diet down-regulates kidney angiotensin-converting enzyme in experimental renal failure. Kidney Int. 2004 Dec;66(6):2155-66. doi: 10.1111/j.1523-1755.2004.66006.x. PMID 15569305
- [Background] Cozzolino M, Staniforth ME, Liapis H, Finch J, Burke SK, Dusso AS, Slatopolsky E. Sevelamer hydrochloride attenuates kidney and cardiovascular calcifications in long-term experimental uremia. Kidney Int. 2003 Nov;64(5):1653-61. doi: 10.1046/j.1523-1755.2003.00284.x. PMID 14531797
- [Background] Taal MW, Roe S, Masud T, Green D, Porter C, Cassidy MJ. Total hip bone mass predicts survival in chronic hemodialysis patients. Kidney Int. 2003 Mar;63(3):1116-20. doi: 10.1046/j.1523-1755.2003.00837.x. PMID 12631095
- [Background] Parfitt AM. Renal bone disease: a new conceptual framework for the interpretation of bone histomorphometry. Curr Opin Nephrol Hypertens. 2003 Jul;12(4):387-403. doi: 10.1097/00041552-200307000-00007. PMID 12815335
- [Background] Riggs BL, Parfitt AM. Drugs used to treat osteoporosis: the critical need for a uniform nomenclature based on their action on bone remodeling. J Bone Miner Res. 2005 Feb;20(2):177-84. doi: 10.1359/JBMR.041114. Epub 2004 Nov 16. PMID 15647810
- [Background] Mansour J, Benyahia M, Harbouche L, Presne C, Moriniere P, Fournier A. Calcimetic AMG 073 at 50 and 100 mg per day. Kidney Int. 2003 Dec;64(6):2324-5. doi: 10.1046/j.1523-1755.2003.341_4.x. No abstract available. PMID 14633162
- [Background] Manns B, Stevens L, Miskulin D, Owen WF Jr, Winkelmayer WC, Tonelli M. A systematic review of sevelamer in ESRD and an analysis of its potential economic impact in Canada and the United States. Kidney Int. 2004 Sep;66(3):1239-47. doi: 10.1111/j.1523-1755.2004.00877.x. PMID 15327423
- [Background] Lacour B, Lucas A, Auchere D, Ruellan N, de Serre Patey NM, Drueke TB. Chronic renal failure is associated with increased tissue deposition of lanthanum after 28-day oral administration. Kidney Int. 2005 Mar;67(3):1062-9. doi: 10.1111/j.1523-1755.2005.00171.x. PMID 15698446
- [Background] Takahashi Y, Tanaka A, Nakamura T, Fukuwatari T, Shibata K, Shimada N, Ebihara I, Koide H. Nicotinamide suppresses hyperphosphatemia in hemodialysis patients. Kidney Int. 2004 Mar;65(3):1099-104. doi: 10.1111/j.1523-1755.2004.00482.x. PMID 14871431
- [Background] Renaud H, Atik A, Herve M, Moriniere P, Hocine C, Belbrik S, Fournier A. Evaluation of vascular calcinosis risk factors in patients on chronic hemodialysis: lack of influence of calcium carbonate. Nephron. 1988;48(1):28-32. doi: 10.1159/000184864. PMID 3340252
- [Background] Wanner C, Krane V, Marz W, Olschewski M, Asmus HG, Kramer W, Kuhn KW, Kutemeyer H, Mann JF, Ruf G, Ritz E; Deutsche Diabetes-Dialyse-Studie (4D) Study Group. Randomized controlled trial on the efficacy and safety of atorvastatin in patients with type 2 diabetes on hemodialysis (4D study): demographic and baseline characteristics. Kidney Blood Press Res. 2004;27(4):259-66. doi: 10.1159/000080241. Epub 2004 Aug 16. PMID 15316128
- [Background] Gale EA, Bingley PJ, Emmett CL, Collier T; European Nicotinamide Diabetes Intervention Trial (ENDIT) Group. European Nicotinamide Diabetes Intervention Trial (ENDIT): a randomised controlled trial of intervention before the onset of type 1 diabetes. Lancet. 2004 Mar 20;363(9413):925-31. doi: 10.1016/S0140-6736(04)15786-3. PMID 15043959
- [Background] Moe SM, Chertow GM, Coburn JW, Quarles LD, Goodman WG, Block GA, Drueke TB, Cunningham J, Sherrard DJ, McCary LC, Olson KA, Turner SA, Martin KJ. Achieving NKF-K/DOQI bone metabolism and disease treatment goals with cinacalcet HCl. Kidney Int. 2005 Feb;67(2):760-71. doi: 10.1111/j.1523-1755.2005.67139.x. PMID 15673327
- [Background] Kauppila LI, Polak JF, Cupples LA, Hannan MT, Kiel DP, Wilson PW. New indices to classify location, severity and progression of calcific lesions in the abdominal aorta: a 25-year follow-up study. Atherosclerosis. 1997 Jul 25;132(2):245-50. doi: 10.1016/s0021-9150(97)00106-8. PMID 9242971
- [Background] Wilson PW, Kauppila LI, O'Donnell CJ, Kiel DP, Hannan M, Polak JM, Cupples LA. Abdominal aortic calcific deposits are an important predictor of vascular morbidity and mortality. Circulation. 2001 Mar 20;103(11):1529-34. doi: 10.1161/01.cir.103.11.1529. PMID 11257080
- [Background] Kiel DP, Kauppila LI, Cupples LA, Hannan MT, O'Donnell CJ, Wilson PW. Bone loss and the progression of abdominal aortic calcification over a 25 year period: the Framingham Heart Study. Calcif Tissue Int. 2001 May;68(5):271-6. doi: 10.1007/BF02390833. PMID 11683533
- [Background] Urena P, Bernard-Poenaru O, Ostertag A, Baudoin C, Cohen-Solal M, Cantor T, de Vernejoul MC. Bone mineral density, biochemical markers and skeletal fractures in haemodialysis patients. Nephrol Dial Transplant. 2003 Nov;18(11):2325-31. doi: 10.1093/ndt/gfg403. PMID 14551361
- [Background] Genant HK, Wu CY, van Kuijk C, Nevitt MC. Vertebral fracture assessment using a semiquantitative technique. J Bone Miner Res. 1993 Sep;8(9):1137-48. doi: 10.1002/jbmr.5650080915. PMID 8237484
- [Background] Grados F, Roux C, de Vernejoul MC, Utard G, Sebert JL, Fardellone P. Comparison of four morphometric definitions and a semiquantitative consensus reading for assessing prevalent vertebral fractures. Osteoporos Int. 2001;12(9):716-22. doi: 10.1007/s001980170046. PMID 11605736
- [Background] Malluche M, Monier-faugère M, wang G, Frazao J, Coburn J, Baker N, McCary LC, Turner JA, Goodman WG: Cinaclacet Hcl reduces bone turn over and bone marrow fibrosa in hemodialysis patients with secondary hyperparathyroidism. ERA XLI congress. AbstractBook Lisboa:P218 (M016), 2004
- [Background] Dament J,Gill M, Confer S, Jones C, Webster J: The bone kinetics of lanthanum in dialysis patient treated with lanthanum carbonate up to 45 years. J Am Soc Nephrol 15 (Abstract):271A (poster FPO 948), 2004
- [Background] Malluche M, Faugère MC, Damment SJP, Webster I: No osteomalacia in dialysis patients treated with lanthanum carbonate up to 4.5 years. J Am Soc Nephrol 15 (supplt Abstract):p270A Poster F P0944,2004
- [Background] De Smet R, Thermote F, Lameire N, Vanholder R: SEVELAMER hydrochloride (Renagel(r)) adsorbs the uremic compounds indoxyl sulfate, indole and p-creso.[Abstract]. J Am Soc Nephrol 15, 2004
- [Background] Block GA, Martin KJ, de Francisco AL, Turner SA, Avram MM, Suranyi MG, Hercz G, Cunningham J, Abu-Alfa AK, Messa P, Coyne DW, Locatelli F, Cohen RM, Evenepoel P, Moe SM, Fournier A, Braun J, McCary LC, Zani VJ, Olson KA, Drueke TB, Goodman WG. Cinacalcet for secondary hyperparathyroidism in patients receiving hemodialysis. N Engl J Med. 2004 Apr 8;350(15):1516-25. doi: 10.1056/NEJMoa031633. PMID 15071126
- [Background] Alsheikh-Ali A, Aboujaily HM, Stanek LJ, coll. e: Increases in HDL cholesterol are the strongest predictions of risk reduction in lipid intervention trials. Circulation 111 (suppltIII):813 Abstract 3754,2004
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086